CLINICAL TRIAL: NCT06602518
Title: Changes in the Sagittal Pharyngeal Airway Dimension Following Leveling and Alignement in Class II Division 2 Patients: A Prospective Clinical Trial
Brief Title: Changes in the Sagittal Pharyngeal Airway Dimension Following Leveling and Alignement in Class II Division 2 Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1/6-2024
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Class II Division 2 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Orthodontics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Levelling and alignment (Experimental)
  Interventions: Procedure: Orthodontic Treatment

INTERVENTIONS:
Procedure: Orthodontic Treatment — All the enrolled patients will undergo conventional fixed appliance therapy by bonding straight wire Roth appliance in the maxillary arch. The bonding procedure will be standardized in all patients and performed by the same operator using light-cured composite. Levelling and alignment will then be started using the following wire sequence: 0.014-in nickel titanium (NiTi), 0.018-in NiTi, 17×25-in Niti, and 19×25-in Niti arch wires. The upper arch will then be stabilized using a 19×25-in stainless steel (SS) arch wire for 2 months. This stage will require approximately 6 months of treatment.

SUMMARY:
Aim of the study: is to compare the changes in the sagittal pharyngeal airway dimension (SPAD) and mandibular position before and after the levelling and alignment stage of orthodontic treatment in Class II division 2 patients.

ELIGIBILITY:
Inclusion Criteria:

* Class II/2 subjects as per the British Standard Institute Classification.
* Age ranging from 12-16 years, with Cervical Vertebral Maturational Index (CVMI) stages 4, and 5.
* Contact between maxillary and mandibular incisors, with the presence of a deep bite of at least 70%.
* Full permanent dentition, aside from the third molars

Exclusion Criteria:

* Previous orthodontic treatment.
* Patients with severe transverse problems, pain and/or clicking sound in the temporomandibular joint (TMJ).
* Patients with craniofacial anomalies or diagnosed syndromes

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the sagittal pharyngeal airway space (SPAD) | 6 months

SECONDARY OUTCOMES:
Changes in the mandibular position | 6 months
Sagittal skeletal measurements | 6 months
Vertical skeletal measurements | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Farah Y Eid, PhD, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Dina Elfouly, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Ahmed Madian, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt